CLINICAL TRIAL: NCT04767893
Title: Evaluation of the Role of sTREM-1 and sUPAR Biomarkers as a Diagnostic Tool and Prognostic Predictor in Sepsis Patients
Brief Title: Diagnostic and Prognostic Biomarkers of Sepsis
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Nahed Fathallah Fahmy, lecturer of medical microbiology & immunology departement -faculty of medicine, Sohag University
Other Study IDs: Soh-Med-21-02-18
Record Dates: First submitted 2021-02-16; First posted 2021-02-23 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Sepsis
Keywords: sTREM-1; sUPAR; CRP
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to evaluate sepsis biomarkers as soluble triggering receptor expressed on myeloid cells 1 (sTREM-1) and soluble urokinase plasminogen activator receptor (sUPAR) in diagnosis of sepsis in comparison to the traditional blood culture and C-reactive protein (CRP) and to evaluate the prognostic value of these biomarkers in comparison to sequential organ failure assessment score (SOFA score), Acute Physiology and Chronic Health Evaluation II ( APACHI score), 28 day mortality.

DETAILED DESCRIPTION:
Sepsis is usually diagnosed in patients have clinically suspected infections with systemic inflammatory response syndrome (SIRS) manifestations. Patients with SIRS as those with trauma or stroke have the same classic infection signs such as fever and elevated leukocytic count, as long as the microbiological diagnosis is the ultimate diagnostic method, but it has poor sensitivity with delayed results. New biomarkers such as sTREM-1 and sUPAR can be used for rapid diagnosis of sepsis and differentiating it from non infectious inflammatory syndromes. Also these soluble biomarkers can be used for predicting the prognosis of sepsis patients

ELIGIBILITY:
Inclusion Criteria:

* Temperature of >38oC
* Heart rate of >90 beats/min
* Respiratory rate of >20 breaths/min
* Partial pressure of arterial carbon dioxide (PaCO2) of <32 mmHg
* White blood cell (WBC) count of >12,000 cells/mm3

Exclusion Criteria:

* HIV patients
* Patients with neutropenia <1000 cells/mm3
* <18 years of age.

Ages: 19 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Our study was conducted on patients admitted to different ICUs in Sohag University Hospital who develop possible clinical signs of sepsis
Sampling Method: Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2019-06-14 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-28 (Actual)

PRIMARY OUTCOMES:
Measurement of the serum level of sTREM-1 (ng/L) in the patients with criteria of SIRS | in the 1st day after appearance of clinical signs of infection
  by ELISA"enzyme linked immunosorbent assay"
Measurement of the serum level of sTREM-1 (ng/L) in the patients with criteria of SIRS | in the 7th day after appearance of clinical signs of infection
  by ELISA"enzyme linked immunosorbent assay"
Measurement of the serum level of sUPAR (ng/L) in the ICU patients | in the 1st day after appearance of clinical signs of infection
  by ELISA"enzyme linked immunosorbent assay"
Measurement of the serum level of sUPAR (ng/L) in the patients with criteria of SIRS | in the 7th day after appearance of clinical signs of infection
  by ELISA"enzyme linked immunosorbent assay"
Measurement of the serum level of CRP (mg/dl) in the patients with criteria of SIRS | in the 1st day after appearance of clinical signs of infection
  by turbidimetry
Measurement of the serum level of CRP (mg/dl) in the patients with criteria of SIRS | in the 7th day after appearance of clinical signs of infection
  by turbidimetry

SECONDARY OUTCOMES:
Acute Physiology and Chronic Health Evaluation II (APACHE II) score designed to measure the severity of disease for adult patients admitted to intensive care units in the with criteria of SIRS | in the 7th day after appearance of clinical signs of infection
  an integer score from 0 to 71
The sequential organ failure assessment score (SOFA score) had been used to determine the extent of organ dysfunction of ICU patients with criteria of SIRS | in the 7th day after appearance of clinical signs of infection
  0-<11

CONTACTS AND LOCATIONS:
Overall Officials: Nahed Fathallah, lecturer, Principal Investigator — Sohag University
Locations (1):
- Faculty of medicine - sohag university, Sohag, Egypt